CLINICAL TRIAL: NCT01713582
Title: A Phase I, Dose-finding Study of the Bromodomain (Brd) Inhibitor OTX015/MK-8628 in Haematological Malignancies
Brief Title: A Dose-finding Study of the Bromodomain (Brd) Inhibitor OTX015/ Birabresib (MK-8628) in Hematologic Malignancies (MK-8628-001)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Oncoethix GmbH, a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 8628-001; OTX015_104 (Other: OncoEthix Protocol Number); 2012-003380-22 (EudraCT Number); MK-8628-001 (Other: Merck Protocol Number); NCT02542358 (obsolete NCT alias)
Record Dates: First submitted 2012-10-22; First posted 2012-10-24 (Estimated); Results first posted 2018-10-01 (Actual); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: Acute Myeloid Leukemia; Diffuse Large B-cell Lymphoma; Acute Lymphoblastic Leukemia; Multiple Myeloma
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Lymphoma, Large B-Cell, Diffuse; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Multiple Myeloma | interventions — OTX015

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (21):
- AL 10 mg QD 14-21 (Experimental): Participants received 10 mg birabresib/OTX015 administered orally (PO), once daily (QD), in a fasted state on Days 1 to 14 of a 21-day cycle.
  Interventions: Drug: OTX015/Birabresib
- AL 20 mg QD 14-21 (Experimental): Participants received 20 mg birabresib/OTX015 administered PO, QD, in a fasted state on Days 1 to 14 of a 21-day cycle.
  Interventions: Drug: OTX015/Birabresib
- AL 40 mg QD 14-21 (Experimental): Participants received 40 mg birabresib/OTX015 administered PO, QD, in a fasted state on Days 1 to 14 of a 21-day cycle.
  Interventions: Drug: OTX015/Birabresib
- AL 20 mg BID 21-21 (Experimental): Participants received 20 mg birabresib/OTX015 administered PO, twice a day (BID), with the first daily dose in a fasted state, on Days 1 to 21 of a 21-day cycle.
  Interventions: Drug: OTX015/Birabresib
- AL 80 mg QD 14-21 (Experimental): Participants received 80 mg birabresib/OTX015 administered PO, QD, in a fasted state on Days 1 to 14 of a 21-day cycle.
  Interventions: Drug: OTX015/Birabresib
- AL 40 mg BID 14-21 (Experimental): Participants received 40 mg birabresib/OTX015 administered PO, twice a day (BID), with the first daily dose in a fasted state, on Days 1 to 14 of a 21-day cycle.
  Interventions: Drug: OTX015/Birabresib
- AL 120 mg QD 14-21 (Experimental): Participants received 120 mg birabresib/OTX015 administered PO, QD, in a fasted state on Days 1 to 14 of a 21-day cycle.
  Interventions: Drug: OTX015/Birabresib
- AL 120 mg QD 21-21 (Experimental): Participants received 120 mg birabresib/OTX015 administered PO, QD, in a fasted state on Days 1 to 21 of a 21-day cycle.
  Interventions: Drug: OTX015/Birabresib
- AL 160 mg QD 14-21 (Experimental): Participants received 160 mg birabresib/OTX015 administered PO, QD, in a fasted state on Days 1 to 14 of a 21-day cycle.
  Interventions: Drug: OTX015/Birabresib
- AML de novo 80 mg QD 14-21 (Experimental): Participants received 80 mg birabresib/OTX015 administered PO, QD, in a fasted state on Days 1 to 14 of a 21-day cycle.
  Interventions: Drug: OTX015/Birabresib
- AML/MDS 80 mg QD 14-21 (Experimental): Participants received 80 mg birabresib/OTX015 administered PO, QD, in a fasted state on Days 1 to 14 of a 21-day cycle.
  Interventions: Drug: OTX015/Birabresib
- OHM 10 mg QD 21-21 (Experimental): Participants received 10 mg birabresib/OTX015 administered PO, QD, in a fasted state on Days 1 to 21 of a 21-day cycle.
  Interventions: Drug: OTX015/Birabresib
- OHM 20 mg QD 21-21 (Experimental): Participants received 20 mg birabresib/OTX015 administered PO, QD, in a fasted state on Days 1 to 21 of a 21-day cycle.
  Interventions: Drug: OTX015/Birabresib
- OHM 40 mg QD 21-21 (Experimental): Participants received 40 mg birabresib/OTX015 administered PO, QD, in a fasted state on Days 1 to 21 of a 21-day cycle.
  Interventions: Drug: OTX015/Birabresib
- OHM 80 mg QD 21-21 (Experimental): Participants received 80 mg birabresib/OTX015 administered PO, QD, in a fasted state on Days 1 to 21 of a 21-day cycle.
  Interventions: Drug: OTX015/Birabresib
- OHM 40 mg BID 21-21 (Experimental): Participants received 40 mg birabresib/OTX015 administered PO, BID, with the first daily dose in a fasted state, on Days 1 to 21 of a 21-day cycle.
  Interventions: Drug: OTX015/Birabresib
- OHM 120 mg QD 21-21 (Experimental): Participants received 120 mg birabresib/OTX015 administered PO, QD, in a fasted state on Days 1 to 21 of a 21-day cycle.
  Interventions: Drug: OTX015/Birabresib
- OHM 120 mg QD 14-21 (Experimental): Participants received 120 mg birabresib/OTX015 administered PO, QD, in a fasted state on Days 1 to 14 of a 21-day cycle.
  Interventions: Drug: OTX015/Birabresib
- OHM 120 mg QD 5-7 (Experimental): Participants received 120 mg birabresib/OTX015 administered PO, QD, in a fasted state on Days 1 to 5 of a 7-day cycle.
  Interventions: Drug: OTX015/Birabresib
- OHM 120 mg QD 7-21 (Experimental): Participants received 120 mg birabresib/OTX015 administered PO, QD, in a fasted state on Days 1 to 7 of a 21-day cycle
  Interventions: Drug: OTX015/Birabresib
- OHM/DLBCL 80 mg QD 14-21 (Experimental): Participants received 80 mg birabresib/OTX015 administered PO, QD, in a fasted state on Days 1 to 14 of a 21-day cycle.
  Interventions: Drug: OTX015/Birabresib

INTERVENTIONS:
Drug: OTX015/Birabresib — OTX015/Birabresib 10 mg, 20 mg, or 40 mg capsules administered orally
  Other Names: MK-8628

SUMMARY:
The primary purpose of this study was to determine the recommended dose (RD) of birabresib (MK-8628) /OTX015 for further phase II studies, in participants with acute leukemia (AL) including acute myeloid leukemia (AML; de novo and secondary to a myelodysplastic syndrome) and acute lymphoblastic leukemia (ALL) or other hematologic malignancies (OHM) including diffuse large B cell lymphoma (DLBCL) and multiple myeloma (MM). The first phase of the study will be a dose escalation phase to determine the Phase II RD using dose-limiting toxicities (DLTs). Once the RD is determined, participants will be enrolled in an expansion phase at the RD to determine preliminary efficacy in AL and OHM cohorts. Participants received therapy in 21-day cycles until disease progression, intolerable toxicity, or treatment interruption for >2 weeks due to toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically proven acute leukemias (AML or ALL) or hematologic malignancies (DLBCL or MM) using standard diagnosis criteria. Acute leukemia includes de novo and secondary to a pre-existing myelodysplastic syndrome, according to the World Health Organization 2008 classification. For DLBCL, an archived formaldehyde-fixed paraffin-embedded block must be available.
* Has failed all standard therapies or for whom standard treatments are contra-indicated:

  * Acute leukemia participants: <60 years old in second relapse or relapsing after allogeneic stem cell transplantation (aSCT) regardless of number of relapses; >60 years old in first relapse with a disease-free interval (DFI) <12 months or further relapse; irrespective of age, in participants relapsing after aSCT, the time elapsed since aSCT should be >90 days; participants with B-cell ALL: Philadelphia chromosome positive (Ph+) must have received ≥2 lines of therapy, including 2 bcr-abl tyrosine-kinase (TK) inhibitors (among imatinib, nilotinib and dasatinib), or only 1 line including 1 TK inhibitor, if the relapse/refractoriness is associated with the detection of a resistance mutation to these inhibitors
  * DLBCL participants: Failed 2 standard lines of therapy (≥1 containing an anti-CD20 monoclonal antibody), or for whom such treatment is contra-indicated
  * MM participants: Adequately exposed to at least one alkylating agent, one corticosteroid, one immunomodulatory drug (IMiD) and bortezomib, or for whom such treatments are contra-indicated.
* For participants with evaluable disease:

  * Advanced leukemia participants must have >5% bone marrow blasts at study entry, without alternative causality (e.g. bone marrow regeneration)
  * DLBCL participants must have ≥1 non-irradiated tumor mass ≥15 mm (long axis of lymph node) or ≥10 mm (short axis of lymph node or extranodal lesions) on spiral computed tomography (CT)-scan.
  * MM participants must have ≥1 of the following: serum monoclonal component >1 g/dL (IgG), or >0.5 g/dL (IgA), or Bence-Jones (BJ) proteinuria >200 mg/24h, or measurable plasmacytoma (not previously irradiated).
* Life expectancy ≥3 months.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2.
* Off previous therapy ≥3 weeks prior to first study drug administration with full recovery from any previous toxicities, except 1) hydroxyurea single agent of in combination (e.g. + 6-Mercaptopurine [6MP]) to control hyperleukocytosis, which should be stopped for ≥48 hours, and 2) rituximab, which should be stopped for ≥3 weeks.
* Recovery from the non-hematologic toxic effects of prior treatment to grade ≤1, according to National Cancer Institute Common Toxicity Criteria (NCI-CTC) classification, except alopecia.
* Adequate bone marrow function.
* Adequate calculated creatinine clearance.
* Adequate liver function tests.
* Complete baseline disease assessment workup prior to first study drug administration.

Exclusion Criteria:

* History of prior malignancy other than those previously treated with a curative intent >3 years ago and without relapse (any tumor) or basal cell skin cancer, in situ cervical cancer, superficial bladder cancer, or high grade intestinal polyps treated adequately, regardless of the DFI.
* Pregnant or lactating women or women of childbearing potential not using adequate contraception. Male participants not using adequate contraception.
* Peripheral cytopenias (i.e. auto-immune hemolytic anemia or thrombocytopenia).
* Acute promyelocytic leukemia or with clinically uncontrolled (i.e. with bleeding) disseminated intravascular coagulation (DIC).
* Chronic graft versus host disease (GVHD) or on immunosuppressive therapy for the control of GVHD.
* Uncontrolled leptomeningeal disease.
* Other tumor location necessitating an urgent therapeutic intervention (palliative care, surgery or radiation therapy), such as spinal cord compression, other compressive mass, uncontrolled painful lesion, bone fracture, etc.
* Unable to swallow oral medications, or has gastrointestinal condition (e.g. malabsorption, resection) deemed to jeopardize intestinal absorption.
* Other serious illness or medical conditions, which, in the investigator's opinion could hamper understanding of the study by the participants, participant's compliance to study treatment, participant's safety or interpretation of study results. These conditions include (but are not restricted to):

  1. Congestive heart failure or angina pectoris except if medically controlled. Previous history of myocardial infarction within 1 year of study entry, uncontrolled hypertension or arrhythmias.
  2. Existence of significant neurologic or psychiatric disorders impairing the ability to obtain consent.
  3. Uncontrolled infection.
  4. Known human immunodeficiency virus (HIV) positivity
* Concurrent treatment with other experimental therapies or participation in another clinical trial within 30 days prior to first study drug administration.
* Concurrent treatment or treatment within 30 days prior to first study drug administration with any other anticancer therapy, except hydroxyurea (+/- 6MP) to control hyperleukocytosis.
* Concomitant treatment with corticosteroids except if chronic treatment with ≤30 mg of methylprednisolone daily or equivalent dose of other corticosteroids.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 141 (Actual)
Dates: Start 2012-12-14 (Actual); Primary Completion 2017-01-20 (Actual); Study Completion 2017-01-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Odore E, Lokiec F, Cvitkovic E, Bekradda M, Herait P, Bourdel F, Kahatt C, Raffoux E, Stathis A, Thieblemont C, Quesnel B, Cunningham D, Riveiro ME, Rezai K. Phase I Population Pharmacokinetic Assessment of the Oral Bromodomain Inhibitor OTX015 in Patients with Haematologic Malignancies. Clin Pharmacokinet. 2016 Mar;55(3):397-405. doi: 10.1007/s40262-015-0327-6. PMID 26341814
- [Derived] Amorim S, Stathis A, Gleeson M, Iyengar S, Magarotto V, Leleu X, Morschhauser F, Karlin L, Broussais F, Rezai K, Herait P, Kahatt C, Lokiec F, Salles G, Facon T, Palumbo A, Cunningham D, Zucca E, Thieblemont C. Bromodomain inhibitor OTX015 in patients with lymphoma or multiple myeloma: a dose-escalation, open-label, pharmacokinetic, phase 1 study. Lancet Haematol. 2016 Apr;3(4):e196-204. doi: 10.1016/S2352-3026(16)00021-1. Epub 2016 Mar 18. PMID 27063978
- [Derived] Berthon C, Raffoux E, Thomas X, Vey N, Gomez-Roca C, Yee K, Taussig DC, Rezai K, Roumier C, Herait P, Kahatt C, Quesnel B, Michallet M, Recher C, Lokiec F, Preudhomme C, Dombret H. Bromodomain inhibitor OTX015 in patients with acute leukaemia: a dose-escalation, phase 1 study. Lancet Haematol. 2016 Apr;3(4):e186-95. doi: 10.1016/S2352-3026(15)00247-1. Epub 2016 Mar 18. PMID 27063977

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 80 participants were enrolled in the acute leukemia (AL) cohort and 78 were treated. 61 participants were enrolled in the other hematological malignancies (OHM) cohort and 60 were treated.
Pre-assignment Details: The study consisted of a dose escalation phase in participants with AL and OHM followed by and expansion phase in 3 cohorts: de novo acute myelocytic leukemia (AML), myelodysplastic syndrome (MDS) AML, and diffuse large B-cell lymphoma (DLBCL).
Groups:
- AL 10 mg QD 14-21: Participants received 10 mg MK-8628/OTX015 administered orally (PO), once daily (QD), in a fasted state on Days 1 to 14 of a 21-day cycle.
- AL 20 mg QD 14-21: Participants received 20 mg MK-8628/OTX015 administered PO, QD, in a fasted state on Days 1 to 14 of a 21-day cycle.
- AL 40 mg QD 14-21: Participants received 40 mg MK-8628/OTX015 administered PO, QD, in a fasted state on Days 1 to 14 of a 21-day cycle.
- AL 20 mg BID 21-21: Participants received 20 mg MK-8628/OTX015 administered PO, twice a day (BID), with the first daily dose in a fasted state, on Days 1 to 21 of a 21-day cycle.
- AL 80 mg QD 14-21; AML de Novo 80 mg QD 14-21; AML/MDS 80 mg QD 14-21; OHM/DLBCL 80 mg QD 14-21: Participants received 80 mg MK-8628/OTX015 administered PO, QD, in a fasted state on Days 1 to 14 of a 21-day cycle.
- AL 40 mg BID 14-21: Participants received 40 mg MK-8628/OTX015 administered PO, twice a day (BID), with the first daily dose in a fasted state, on Days 1 to 14 of a 21-day cycle.
- AL 120 mg QD 14-21; OHM 120 mg QD 14-21: Participants received 120 mg MK-8628/OTX015 administered PO, QD, in a fasted state on Days 1 to 14 of a 21-day cycle.
- AL 120 mg QD 21-21; OHM 120 mg QD 21-21: Participants received 120 mg MK-8628/OTX015 administered PO, QD, in a fasted state on Days 1 to 21 of a 21-day cycle.
- AL 160 mg QD 14-21: Participants received 160 mg MK-8628/OTX015 administered PO, QD, in a fasted state on Days 1 to 14 of a 21-day cycle.
- OHM 10 mg QD 21-21: Participants received 10 mg MK-8628/OTX015 administered PO, QD, in a fasted state on Days 1 to 21 of a 21-day cycle.
- OHM 20 mg QD 21-21: Participants received 20 mg MK-8628/OTX015 administered PO, QD, in a fasted state on Days 1 to 21 of a 21-day cycle.
- OHM 40 mg QD 21-21: Participants received 40 mg MK-8628/OTX015 administered PO, QD, in a fasted state on Days 1 to 21 of a 21-day cycle.
- OHM 80 mg QD 21-21: Participants received 80 mg MK-8628/OTX015 administered PO, QD, in a fasted state on Days 1 to 21 of a 21-day cycle.
- OHM 40 mg BID 21-21: Participants received 40 mg MK-8628/OTX015 administered PO, BID, with the first daily dose in a fasted state, on Days 1 to 21 of a 21-day cycle.
- OHM 120 mg QD 5-7: Participants received 120 mg MK-8628/OTX015 administered PO, QD, in a fasted state on Days 1 to 5 of a 7-day cycle.
- OHM 120 mg QD 7-21: Participants received 120 mg MK-8628/OTX015 administered PO, QD, in a fasted state on Days 1 to 7 of a 21-day cycle.
Period: Overall Study
Arm/Group | AL 10 mg QD 14-21 | AL 20 mg QD 14-21 | AL 40 mg QD 14-21 | AL 20 mg BID 21-21 | AL 80 mg QD 14-21 | AL 40 mg BID 14-21 | AL 120 mg QD 14-21 | AL 120 mg QD 21-21 | AL 160 mg QD 14-21 | AML de Novo 80 mg QD 14-21 | AML/MDS 80 mg QD 14-21 | OHM 10 mg QD 21-21 | OHM 20 mg QD 21-21 | OHM 40 mg QD 21-21 | OHM 80 mg QD 21-21 | OHM 40 mg BID 21-21 | OHM 120 mg QD 21-21 | OHM 120 mg QD 14-21 | OHM 120 mg QD 5-7 | OHM 120 mg QD 7-21 | OHM/DLBCL 80 mg QD 14-21
Started | 3 (Number treated) | 3 (Number treated) | 4 (Number treated) | 3 (Number treated) | 4 (Number treated) | 8 (Number treated) | 7 (Number treated) | 6 (Number treated) | 6 (Number treated) | 18 (Number treated) | 16 (Number treated) | 5 (Number treated) | 3 (Number treated) | 4 (Number treated) | 7 (Number treated) | 6 (Number treated) | 7 (Number treated) | 3 (Number treated) | 5 (Number treated) | 5 (Number treated) | 15 (Number treated)
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 3 | 3 | 4 | 3 | 4 | 8 | 7 | 6 | 6 | 18 | 16 | 5 | 3 | 4 | 7 | 6 | 7 | 3 | 5 | 5 | 15
Not completed — Disease progression | 3 | 3 | 3 | 2 | 3 | 3 | 3 | 3 | 3 | 11 | 10 | 5 | 3 | 3 | 6 | 6 | 5 | 2 | 3 | 5 | 15
Not completed — Death | 0 | 0 | 0 | 1 | 1 | 3 | 3 | 2 | 3 | 4 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse event-related | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Adverse event-unrelated | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal of consent | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Stopped to receive bone marrow graft | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Disease progression and adverse event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AL 10 mg QD 14-21 | AL 20 mg QD 14-21 | AL 40 mg QD 14-21 | AL 20 mg BID 21-21 | AL 80 mg QD 14-21 | AL 40 mg BID 14-21 | AL 120 mg QD 14-21 | AL 120 mg QD 21-21 | AL 160 mg QD 14-21 | AML de Novo 80 mg QD 14-21 | AML/MDS 80 mg QD 14-21 | OHM 10 mg QD 21-21 | OHM 20 mg QD 21-21 | OHM 40 mg QD 21-21 | OHM 80 mg QD 21-21 | OHM 40 mg BID 21-21 | OHM 120 mg QD 21-21 | OHM 120 mg QD 14-21 | OHM 120 mg QD 5-7 | OHM 120 mg QD 7-21 | OHM/DLBCL 80 mg QD 14-21 | Total
Number analyzed (Participants) | 3 | 3 | 4 | 3 | 4 | 8 | 7 | 6 | 6 | 18 | 16 | 5 | 3 | 4 | 7 | 6 | 7 | 3 | 5 | 5 | 15 | 138
Age, Continuous [Mean (Standard Deviation); unit: Years] | 67.0 (3.5) [65.0 to 71.0] | 54.7 (19.6) [32.0 to 66.0] | 73.8 (2.1) [71.0 to 76.0] | 77.7 (2.3) [75.0 to 79.0] | 70.0 (10.6) [55.0 to 80.0] | 65.8 (16.3) [33.0 to 85.0] | 65.3 (13.9) [42.0 to 79.0] | 58.5 (24.1) [19.0 to 80.0] | 57.8 (16.6) [26.0 to 75.0] | 65.6 (10.0) [45.0 to 79.0] | 67.2 (8.2) [48.0 to 81.0] | 65.2 (15.5) | 74.7 (7.4) | 69.0 (8.4) | 59.4 (18.5) | 54.7 (13.0) | 55.6 (19.3) | 66.0 (13.2) | 62.4 (8.4) | 66.8 (8.3) | 58.5 (14.1) | 63.7 (13.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 2 | 1 | 0 | 3 | 3 | 2 | 0 | 8 | 3 | 0 | 1 | 2 | 3 | 3 | 2 | 0 | 0 | 5 | 4 | 46
  Male | 2 | 0 | 2 | 2 | 4 | 5 | 4 | 4 | 6 | 10 | 13 | 5 | 2 | 2 | 4 | 3 | 5 | 3 | 5 | 0 | 11 | 92
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicities (DLTs)
Description: A DLT was graded using the National Cancer Institute-Common Toxicity Criteria for Adverse Events (NCI-CTCAE) version 4.02 and defined as any of the following: grade 3 or 4 non-hematologic adverse events unless they were not optimally treated with supportive care; grade 3 or 4 asymptomatic laboratory abnormal values lasting >7 days; prolonged grade 2 toxicity (lasting more than 2 weeks) leading to treatment interruption and/or dose reduction; pancytopenia with a hypocellular bone marrow and no marrow blasts lasting ≥6 weeks (AL participants); grade 3 neutropenia with fever or infection (OHM participants); grade 3 thrombocytopenia with bleeding (OHM participants); or grade 4 neutropenia or thrombocytopenia, regardless of symptoms and lasting ≥3 days (OHM participants).
Time Frame: Cycle 1 (Up to 21 days)
Population: All participants who received at least 85% of the intended dose of study therapy during the first cycle (i.e. >12 days at full dose for AL and >18 days at full dose for other hematological malignancies) or discontinued from the study due to a DLT attributable to study therapy.
Measure: Count of Participants; unit: Participants
Groups:
- AL 40 mg BID 14-21: Participants received 40 mg MK-8628/OTX015 administered PO, BID, with the first daily dose in a fasted state, on Days 1 to 14 of a 21-day cycle.
Arm/Group | AL 10 mg QD 14-21 | AL 20 mg QD 14-21 | AL 40 mg QD 14-21 | AL 20 mg BID 21-21 | AL 80 mg QD 14-21 | AL 40 mg BID 14-21 | AL 120 mg QD 14-21 | AL 120 mg QD 21-21 | AL 160 mg QD 14-21 | AML de Novo 80 mg QD 14-21 | AML/MDS 80 mg QD 14-21 | OHM 10 mg QD 21-21 | OHM 20 mg QD 21-21 | OHM 40 mg QD 21-21 | OHM 80 mg QD 21-21 | OHM 40 mg BID 21-21 | OHM 120 mg QD 21-21 | OHM 120 mg QD 14-21 | OHM 120 mg QD 5-7 | OHM 120 mg QD 7-21 | OHM/DLBCL 80 mg QD 14-21
Number analyzed (Participants) | 3 | 3 | 4 | 3 | 4 | 6 | 6 | 6 | 6 | 17 | 14 | 3 | 3 | 3 | 7 | 6 | 6 | 3 | 4 | 5 | 14
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 2 | 5 | 4 | 2 | 3 | 2 | 0

2. Secondary Outcome: Number of Participants Who Experienced at Least One Adverse Event (AE)
Description: AE was defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which did not necessarily have to have a causal relationship with this treatment. An AE could therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product/protocol specified procedure, whether or not considered related to the medicinal product/protocol specified procedure. Any worsening of a preexisting condition temporally associated with the use of the product was also an AE. AEs were collected during the entire time frame of treatment plus up to 40 days of follow-up.
Time Frame: Up to 40 days after last dose of study therapy (Up to 28 months)
Population: All participants who received at least one dose of study therapy.
Measure: Count of Participants; unit: Participants
Groups:
- AL 10 mg QD 14-21: Participants received 10 mg MK-8628/OTX015 administered PO, QD, in a fasted state on Days 1 to 14 of a 21-day cycle.
- AL 20 mg BID 21-21: Participants received 20 mg MK-8628/OTX015 administered PO, BID, with the first daily dose in a fasted state, on Days 1 to 21 of a 21-day cycle.
Arm/Group | AL 10 mg QD 14-21 | AL 20 mg QD 14-21 | AL 40 mg QD 14-21 | AL 20 mg BID 21-21 | AL 80 mg QD 14-21 | AL 40 mg BID 14-21 | AL 120 mg QD 14-21 | AL 120 mg QD 21-21 | AL 160 mg QD 14-21 | AML de Novo 80 mg QD 14-21 | AML/MDS 80 mg QD 14-21 | OHM 10 mg QD 21-21 | OHM 20 mg QD 21-21 | OHM 40 mg QD 21-21 | OHM 80 mg QD 21-21 | OHM 40 mg BID 21-21 | OHM 120 mg QD 21-21 | OHM 120 mg QD 14-21 | OHM 120 mg QD 5-7 | OHM 120 mg QD 7-21 | OHM/DLBCL 80 mg QD 14-21
Number analyzed (Participants) | 3 | 3 | 4 | 3 | 4 | 8 | 7 | 6 | 6 | 18 | 16 | 5 | 3 | 4 | 7 | 6 | 7 | 3 | 5 | 5 | 15
Participants | 3 | 3 | 4 | 3 | 4 | 8 | 7 | 6 | 6 | 18 | 16 | 5 | 3 | 4 | 7 | 6 | 7 | 3 | 5 | 5 | 15

3. Secondary Outcome: Number of Participants Who Discontinued Study Therapy Due to AEs
Description: All participants who discontinued study therapy due to an AE at any time during treatment.
Time Frame: From time of first dose of study therapy until the end of treatment (up to 26 months)
Population: All participants who received at least one dose of study therapy.
Measure: Count of Participants; unit: Participants
Arm/Group | AL 10 mg QD 14-21 | AL 20 mg QD 14-21 | AL 40 mg QD 14-21 | AL 20 mg BID 21-21 | AL 80 mg QD 14-21 | AL 40 mg BID 14-21 | AL 120 mg QD 14-21 | AL 120 mg QD 21-21 | AL 160 mg QD 14-21 | AML de Novo 80 mg QD 14-21 | AML/MDS 80 mg QD 14-21 | OHM 10 mg QD 21-21 | OHM 20 mg QD 21-21 | OHM 40 mg QD 21-21 | OHM 80 mg QD 21-21 | OHM 40 mg BID 21-21 | OHM 120 mg QD 21-21 | OHM 120 mg QD 14-21 | OHM 120 mg QD 5-7 | OHM 120 mg QD 7-21 | OHM/DLBCL 80 mg QD 14-21
Number analyzed (Participants) | 3 | 3 | 4 | 3 | 4 | 8 | 7 | 6 | 6 | 18 | 16 | 5 | 3 | 4 | 7 | 6 | 7 | 3 | 5 | 5 | 15
Participants | 0 | 0 | 1 | 1 | 1 | 3 | 2 | 2 | 4 | 7 | 4 | 0 | 0 | 1 | 1 | 1 | 2 | 1 | 2 | 0 | 0

4. Secondary Outcome: Number of Participants Whose Best Response Was Partial Response (PR) or Complete Response (CR)
Description: Best response was determined from the start of treatment until disease progression, recurrence, or completion of 26 months of treatment. Partial and complete response was assessed by bone marrow aspiration (AL participants); or computed tomography scan, magnetic resonance imaging, positron emission tomography, or X-ray (OHM participants) using standard criteria. Acute leukemia participants were assessed based on the recommendations from the European LeukemiaNet Döhner 2010); lymphoma participants according to Cheson 2007; and MM participants according to Durie 2006.
Time Frame: From time of first dose of study therapy until the end of treatment (up to 26 months)
Population: All participants who received one dose of study therapy and had at least one available tumor assessment by the end of Cycle 2 or later or with earlier evidence of response or progression.
Measure: Number; unit: Participants
Arm/Group | AL 10 mg QD 14-21 | AL 20 mg QD 14-21 | AL 40 mg QD 14-21 | AL 20 mg BID 21-21 | AL 80 mg QD 14-21 | AL 40 mg BID 14-21 | AL 120 mg QD 14-21 | AL 120 mg QD 21-21 | AL 160 mg QD 14-21 | AML de Novo 80 mg QD 14-21 | AML/MDS 80 mg QD 14-21 | OHM 10 mg QD 21-21 | OHM 20 mg QD 21-21 | OHM 40 mg QD 21-21 | OHM 80 mg QD 21-21 | OHM 40 mg BID 21-21 | OHM 120 mg QD 21-21 | OHM 120 mg QD 14-21 | OHM 120 mg QD 5-7 | OHM 120 mg QD 7-21 | OHM/DLBCL 80 mg QD 14-21
Number analyzed (Participants) | 3 | 3 | 4 | 3 | 4 | 8 | 7 | 6 | 6 | 18 | 16 | 5 | 3 | 4 | 7 | 6 | 7 | 3 | 5 | 5 | 15
Participants | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 1

5. Secondary Outcome: Maximum Concentration (Cmax) of MK-8628/OTX015
Description: Data were collected in Cycle 1 according to dosing regimen and enrollment position at the following sampling schedules: 1) Complete QD for the first 3 participants per dose level: Pre-infusion and 1, 4, 8, 12, and 24 hours (h) + 1 sampling at either 10h or 16h post-infusion on Days 1 and 2 and on Days 8, 15, and 22 pre-infusion per dose level; 2) Limited QD for participants 4 and higher: Pre-infusion and 1, 4, 6, and 8h post-infusion on Days 1 and 2 and on Days 8, 15, and 22 pre-infusion per dose level; 3) BID: Pre-infusion and at 20 minutes and 1, 2.25, 3.25. 9, 12, and 24h post-infusion on Days 1 and 2 and on Days 8, 15, and 22 pre-infusion per dose level.
  Blood samples for Cmax were measured using liquid chromatography-tandem mass spectrometry and analyzed using a nonlinear mixed-effects modelling software program Monolix version 4.3.2. Results for each dose level and method of administration included participants from both AL and OHM cohorts and different regimen frequencies.
Time Frame: Cycle 1: Pre-infusion and 20 minutes; 1, 2.25, 3.25, 4, 6, 8, 9, 12, and 24 hours plus one sampling at either 10 hour or 16 hour post-infusion on Days 1 and 2 and on Days 8, 15, and 22 pre-infusion dependent on dose regimen and enrollment position
Population: All participants that received at least 1 dose of study therapy and had evaluable data for endpoint. Results were pooled by dose taken and not by disease or regimen.
Measure: Mean (Standard Deviation); unit: ug/L
Groups:
- 10 mg QD Dose Escalation Cohort: Participants received 10 mg MK-8628/OTX015 administered PO, QD, in a fasted state.
- 20 mg QD Dose Escalation Cohort: Participants received 20 mg MK-8628/OTX015 administered PO, QD, in a fasted state.
- 40 mg QD Dose Escalation Cohort: Participants received 40 mg MK-8628/OTX015 administered PO, QD, in a fasted state.
- 20 mg BID Dose Escalation Cohort: Participants received 20 mg MK-8628/OTX015 administered PO, BID, with the first daily dose in a fasted state.
- 80 mg QD Dose Escalation Cohort; 80 mg QD Expansion Cohort: Participants received 80 mg MK-8628/OTX015 administered PO, QD, in a fasted state.
- 40 mg BID Dose Escalation Cohort: Participants received 40 mg MK-8628/OTX015 administered PO, BID, with the first daily dose in a fasted state.
- 120 mg QD Dose Escalation Cohort: Participants received 120 mg MK-8628/OTX015 administered PO, QD, in a fasted state.
- 160 mg QD Dose Escalation Cohort: Participants received 160 mg MK-8628/OTX015 administered PO, QD, in a fasted state.
Arm/Group | 10 mg QD Dose Escalation Cohort | 20 mg QD Dose Escalation Cohort | 40 mg QD Dose Escalation Cohort | 20 mg BID Dose Escalation Cohort | 80 mg QD Dose Escalation Cohort | 40 mg BID Dose Escalation Cohort | 120 mg QD Dose Escalation Cohort | 160 mg QD Dose Escalation Cohort | 80 mg QD Expansion Cohort
Number analyzed (Participants) | 8 | 6 | 8 | 3 | 11 | 13 | 31 | 5 | 49
ug/L | 131 (56.5) | 275 (104) | 627 (328) | 453 (185) | 1131 (650) | 556 (194) | 1425 (555) | 1292 (572) | 982 (316)

6. Secondary Outcome: Time to Maximum Concentration (Tmax) of MK-8628/OTX015
Description: Data were collected in Cycle 1 according to dosing regimen and enrollment position at the following sampling schedules: 1) Complete QD for the first 3 participants per dose level: Pre-infusion and 1, 4, 8, 12, and 24h + 1 sampling at either 10h or 16h post-infusion on Days 1 and 2 and on Days 8, 15, and 22 pre-infusion per dose level; 2) Limited QD for participants 4 and higher: Pre-infusion and 1, 4, 6, and 8h post-infusion on Days 1 and 2 and on Days 8, 15, and 22 pre-infusion per dose level; 3) BID: Pre-infusion and at 20 minutes and 1, 2.25, 3.25. 9, 12, and 24h post-infusion on Days 1 and 2 and on Days 8, 15, and 22 pre-infusion per dose level.
  Blood samples for Tmax were measured using liquid chromatography-tandem mass spectrometry and analyzed using a nonlinear mixed-effects modelling software program Monolix version 4.3.2. Results for each dose level and method of administration included participants from both AL and OHM cohorts and different regimen frequencies.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | 10 mg QD Dose Escalation Cohort | 20 mg QD Dose Escalation Cohort | 40 mg QD Dose Escalation Cohort | 20 mg BID Dose Escalation Cohort | 80 mg QD Dose Escalation Cohort | 40 mg BID Dose Escalation Cohort | 120 mg QD Dose Escalation Cohort | 160 mg QD Dose Escalation Cohort | 80 mg QD Expansion Cohort
Number analyzed (Participants) | 8 | 6 | 8 | 3 | 11 | 13 | 31 | 5 | 49
Hours | 1.78 (1.37) | 3.03 (1.54) | 1.75 (1.04) | 1.92 (0.795) | 3.44 (1.21) | 2.73 (2.08) | 3.48 (1.35) | 4.22 (2.46) | 3.07 (1.79)

7. Secondary Outcome: Apparent Terminal Half-Life (t1/2) of MK-8628/OTX015
Description: Data were collected in Cycle 1 according to dosing regimen and enrollment position at the following sampling schedules: 1) Complete QD for the first 3 participants per dose level: Pre-infusion and 1, 4, 8, 12, and 24h + 1 sampling at either 10h or 16h post-infusion on Days 1 and 2 and on Days 8, 15, and 22 pre-infusion per dose level; 2) Limited QD for participants 4 and higher: Pre-infusion and 1, 4, 6, and 8h post-infusion on Days 1 and 2 and on Days 8, 15, and 22 pre-infusion per dose level; 3) BID: Pre-infusion and at 20 minutes and 1, 2.25, 3.25. 9, 12, and 24h post-infusion on Days 1 and 2 and on Days 8, 15, and 22 pre-infusion per dose level.
  Blood samples for t1/2 were measured using liquid chromatography-tandem mass spectrometry and analyzed using a nonlinear mixed-effects modelling software program Monolix version 4.3.2. Results for each dose level and method of administration included participants from both AL and OHM cohorts and different regimen frequencies.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Hours
Groups:
- 10 mg QD Dose Escalation Cohort: Participants received 10 mg MK-8628/OTX015 administered PO, QD in a fasted state.
Arm/Group | 10 mg QD Dose Escalation Cohort | 20 mg QD Dose Escalation Cohort | 40 mg QD Dose Escalation Cohort | 20 mg BID Dose Escalation Cohort | 80 mg QD Dose Escalation Cohort | 40 mg BID Dose Escalation Cohort | 120 mg QD Dose Escalation Cohort | 160 mg QD Dose Escalation Cohort | 80 mg QD Expansion Cohort
Number analyzed (Participants) | 8 | 6 | 8 | 3 | 11 | 13 | 31 | 5 | 49
Hours | 3.65 (0.695) | 4.78 (1.53) | 4.55 (0.533) | 4.71 (1.1) | 4.62 (0.673) | 4.70 (1.19) | 4.49 (1.01) | 3.87 (0.712) | 4.27 (0.940)

8. Secondary Outcome: Area Under the Concentration Time Curve of MK-8628/OTX015 From Time 0 to Infinity (AUC 0-inf)
Description: Data were collected in Cycle 1 according to dosing regimen and enrollment position at the following sampling schedules: 1) Complete QD for the first 3 participants per dose level: Pre-infusion and 1, 4, 8, 12, and 24h + 1 sampling at either 10h or 16h post-infusion on Days 1 and 2 and on Days 8, 15, and 22 pre-infusion per dose level; 2) Limited QD for participants 4 and higher: Pre-infusion and 1, 4, 6, and 8h post-infusion on Days 1 and 2 and on Days 8, 15, and 22 pre-infusion per dose level; 3) BID: Pre-infusion and at 20 minutes and 1, 2.25, 3.25. 9, 12, and 24h post-infusion on Days 1 and 2 and on Days 8, 15, and 22 pre-infusion per dose level.
  Blood samples for AUC 0-first were measured using liquid chromatography-tandem mass spectrometry and analyzed using a nonlinear mixed-effects modelling software program Monolix version 4.3.2. Results for each dose level and method of administration included participants from both AL and OHM cohorts and different regimen frequencies.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | 10 mg QD Dose Escalation Cohort | 20 mg QD Dose Escalation Cohort | 40 mg QD Dose Escalation Cohort | 20 mg BID Dose Escalation Cohort | 80 mg QD Dose Escalation Cohort | 40 mg BID Dose Escalation Cohort | 120 mg QD Dose Escalation Cohort | 160 mg QD Dose Escalation Cohort | 80 mg QD Expansion Cohort
Number analyzed (Participants) | 8 | 6 | 8 | 3 | 11 | 13 | 31 | 5 | 49
hr*ng/mL | 1060 (191) | 2828 (983) | 5301 (924) | 3947 (1184) | 11910 (6987) | 5619 (1895) | 15240 (6021) | 13190 (3183) | 9833 (2968)

9. Secondary Outcome: Apparent Total Body Clearance (CL/F) of MK-8628/OTX015
Description: Data were collected in Cycle 1 according to dosing regimen and enrollment position at the following sampling schedules: 1) Complete QD for the first 3 participants per dose level: Pre-infusion and 1, 4, 8, 12, and 24h + 1 sampling at either 10h or 16h post-infusion on Days 1 and 2 and on Days 8, 15, and 22 pre-infusion per dose level; 2) Limited QD for participants 4 and higher: Pre-infusion and 1, 4, 6, and 8h post-infusion on Days 1 and 2 and on Days 8, 15, and 22 pre-infusion per dose level; 3) BID: Pre-infusion and at 20 minutes and 1, 2.25, 3.25. 9, 12, and 24h post-infusion on Days 1 and 2 and on Days 8, 15, and 22 pre-infusion per dose level.
  Blood samples for CL/F were measured using liquid chromatography-tandem mass spectrometry and analyzed using a nonlinear mixed-effects modelling software program Monolix version 4.3.2. Results for each dose level and method of administration included participants from both AL and OHM cohorts and different regimen frequencies.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: L/hour
Arm/Group | 10 mg QD Dose Escalation Cohort | 20 mg QD Dose Escalation Cohort | 40 mg QD Dose Escalation Cohort | 20 mg BID Dose Escalation Cohort | 80 mg QD Dose Escalation Cohort | 40 mg BID Dose Escalation Cohort | 120 mg QD Dose Escalation Cohort | 160 mg QD Dose Escalation Cohort | 80 mg QD Expansion Cohort
Number analyzed (Participants) | 8 | 6 | 8 | 3 | 11 | 13 | 31 | 5 | 49
L/hour | 9.71 (1.73) | 7.67 (2.13) | 7.76 (1.38) | 6.53 (1.88) | 7.91 (3.04) | 7.49 (2.18) | 8.61 (2.22) | 12.7 (2.80) | 8.87 (2.60)

10. Secondary Outcome: Volume of Distribution at Steady State (Vz/F) of MK-8628/OTX015
Description: Data were collected in Cycle 1 according to dosing regimen and enrollment position at the following sampling schedules: 1) Complete QD for the first 3 participants per dose level: Pre-infusion and 1, 4, 8, 12, and 24h + 1 sampling at either 10h or 16h post-infusion on Days 1 and 2 and on Days 8, 15, and 22 pre-infusion per dose level; 2) Limited QD for participants 4 and higher: Pre-infusion and 1, 4, 6, and 8h post-infusion on Days 1 and 2 and on Days 8, 15, and 22 pre-infusion per dose level; 3) BID: Pre-infusion and at 20 minutes and 1, 2.25, 3.25. 9, 12, and 24h post-infusion on Days 1 and 2 and on Days 8, 15, and 22 pre-infusion per dose level.
  Blood samples for Vz/F were measured using liquid chromatography-tandem mass spectrometry and analyzed using a nonlinear mixed-effects modelling software program Monolix version 4.3.2. Results for each dose level and method of administration included participants from both AL and OHM cohorts and different regimen frequencies.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | 10 mg QD Dose Escalation Cohort | 20 mg QD Dose Escalation Cohort | 40 mg QD Dose Escalation Cohort | 20 mg BID Dose Escalation Cohort | 80 mg QD Dose Escalation Cohort | 40 mg BID Dose Escalation Cohort | 120 mg QD Dose Escalation Cohort | 160 mg QD Dose Escalation Cohort | 80 mg QD Expansion Cohort
Number analyzed (Participants) | 8 | 6 | 8 | 3 | 11 | 13 | 31 | 5 | 49
Liters | 49.6 (1.0) | 49.1 (3.51) | 50.8 (10.0) | 42.4 (4.25) | 50.4 (17.5) | 48.2 (9.22) | 54.2 (14.4) | 69.3 (13.3) | 52.0 (9.18)

ADVERSE EVENTS:
Time Frame: Adverse events were monitored up to 40 days after last dose of study therapy (Up to 28 months).
Description: The safety population consisted of all participants who received at least one dose of study therapy.
Arm/Group | AL 10 mg QD 14-21 | AL 20 mg QD 14-21 | AL 40 mg QD 14-21 | AL 20 mg BID 21-21 | AL 80 mg QD 14-21 | AL 40 mg BID 14-21 | AL 120 mg QD 14-21 | AL 120 mg QD 21-21 | AL 160 mg QD 14-21 | AML de Novo 80 mg QD 14-21 | AML/MDS 80 mg QD 14-21 | OHM 10 mg QD 21-21 | OHM 20 mg QD 21-21 | OHM 40 mg QD 21-21 | OHM 40 mg BID 21-21 | OHM 120 mg QD 21-21 | OHM 120 mg QD 14-21 | OHM 120 mg QD 5-7 | OHM 120 mg QD 7-21 | OHM/DLBCL 80 mg QD 14-21 | OHM 80 mg QD 21-21
All-Cause Mortality (participants affected / at risk) | 3/3 | 3/3 | 4/4 | 3/3 | 4/4 | 7/8 | 7/7 | 6/6 | 6/6 | 15/18 | 15/16 | 3/5 | 2/3 | 2/4 | 4/6 | 5/7 | 1/3 | 2/5 | 5/5 | 9/15 | 4/7
Serious Adverse Events (participants affected / at risk) | 1/3 | 2/3 | 3/4 | 1/3 | 3/4 | 7/8 | 6/7 | 5/6 | 4/6 | 14/18 | 14/16 | 3/5 | 1/3 | 0/4 | 5/6 | 6/7 | 2/3 | 2/5 | 2/5 | 5/15 | 4/7
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 4/4 | 3/3 | 4/4 | 8/8 | 7/7 | 6/6 | 6/6 | 18/18 | 16/16 | 5/5 | 3/3 | 4/4 | 6/6 | 7/7 | 3/3 | 5/5 | 5/5 | 15/15 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AL 10 mg QD 14-21 (N=3) | AL 20 mg QD 14-21 (N=3) | AL 40 mg QD 14-21 (N=4) | AL 20 mg BID 21-21 (N=3) | AL 80 mg QD 14-21 (N=4) | AL 40 mg BID 14-21 (N=8) | AL 120 mg QD 14-21 (N=7) | AL 120 mg QD 21-21 (N=6) | AL 160 mg QD 14-21 (N=6) | AML de Novo 80 mg QD 14-21 (N=18) | AML/MDS 80 mg QD 14-21 (N=16) | OHM 10 mg QD 21-21 (N=5) | OHM 20 mg QD 21-21 (N=3) | OHM 40 mg QD 21-21 (N=4) | OHM 40 mg BID 21-21 (N=6) | OHM 120 mg QD 21-21 (N=7) | OHM 120 mg QD 14-21 (N=3) | OHM 120 mg QD 5-7 (N=5) | OHM 120 mg QD 7-21 (N=5) | OHM/DLBCL 80 mg QD 14-21 (N=15) | OHM 80 mg QD 21-21 (N=7)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 3 | 1 | 1 | 2 | 1 | 2 | 1 | 4 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhagic disorder (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 1 | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 5 | 2 | 1 | 1 | 1 | 0 | 2
Atrial flutter (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1
Anorectal disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 2 | 1 | 0
Faecal incontinence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Disease progression (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
General physical health deterioration (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Puncture site haemorrhage (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Aspergillosis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchopulmonary aspergillosis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cerebral aspergillosis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Device related infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Enterobacter infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infectious peritonitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lung infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lung infection pseudomonal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neutropenic sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pseudomonas infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0 | 3 | 1 | 0 | 3 | 5 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Septic shock (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Viral skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood calcium increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Enterococcus test positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Factor VII deficiency (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperbilirubinaemia (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Transaminases increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Convulsion (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Depressed level of consciousness (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhage intracranial (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oliguria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Bronchial haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Chest pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Air embolism (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AL 10 mg QD 14-21 (N=3) | AL 20 mg QD 14-21 (N=3) | AL 40 mg QD 14-21 (N=4) | AL 20 mg BID 21-21 (N=3) | AL 80 mg QD 14-21 (N=4) | AL 40 mg BID 14-21 (N=8) | AL 120 mg QD 14-21 (N=7) | AL 120 mg QD 21-21 (N=6) | AL 160 mg QD 14-21 (N=6) | AML de Novo 80 mg QD 14-21 (N=18) | AML/MDS 80 mg QD 14-21 (N=16) | OHM 10 mg QD 21-21 (N=5) | OHM 20 mg QD 21-21 (N=3) | OHM 40 mg QD 21-21 (N=4) | OHM 40 mg BID 21-21 (N=6) | OHM 120 mg QD 21-21 (N=7) | OHM 120 mg QD 14-21 (N=3) | OHM 120 mg QD 5-7 (N=5) | OHM 120 mg QD 7-21 (N=5) | OHM/DLBCL 80 mg QD 14-21 (N=15) | OHM 80 mg QD 21-21 (N=7)
Anaemia (Blood and lymphatic system disorders) | 2 | 2 | 3 | 1 | 4 | 7 | 5 | 5 | 3 | 9 | 7 | 1 | 0 | 1 | 3 | 1 | 1 | 3 | 0 | 1 | 4
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 0 | 1 | 0 | 1 | 2 | 1 | 2 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhagic disorder (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 1 | 2 | 2 | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 1 | 1 | 1 | 0 | 2 | 0 | 2 | 0 | 1 | 7 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lymph node pain (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 1 | 1 | 1
Splenomegaly (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 2 | 2 | 0 | 3 | 6 | 2 | 2 | 2 | 7 | 3 | 0 | 0 | 2 | 1 | 3 | 1 | 2 | 0 | 4 | 3
Arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Conduction disorder (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Supraventricular extrasystoles (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Factor V deficiency (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Deafness (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Conjunctival haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctivitis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dry eye (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Exophthalmos (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Eye disorder (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye pain (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Periorbital oedema (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Photophobia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ulcerative keratitis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Visual acuity reduced (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 1 | 4 | 2 | 1 | 1 | 4 | 0 | 2 | 0 | 0 | 1 | 2 | 0 | 1 | 3 | 0 | 1
Anorectal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Breath odour (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cheilitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 2 | 5 | 3 | 0 | 1 | 1 | 1 | 3 | 0 | 0 | 2 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 4 | 4 | 4 | 6 | 4 | 9 | 11 | 0 | 0 | 3 | 4 | 5 | 2 | 4 | 3 | 9 | 6
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 2 | 1 | 0 | 1 | 1 | 5 | 2
Duodenogastric reflux (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 2 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Faecal incontinence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Faeces discoloured (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1
Gingival bleeding (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gingival disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gingival hypertrophy (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gingival pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1
Melaena (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mouth haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 2 | 4 | 2 | 3 | 3 | 7 | 11 | 0 | 0 | 1 | 3 | 2 | 1 | 4 | 4 | 7 | 3
Odynophagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oral pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 1 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1
Tongue coated (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 2 | 1 | 1 | 1 | 3 | 3 | 0 | 0 | 2 | 3 | 3 | 0 | 1 | 2 | 2 | 0
Asthenia (General disorders) | 1 | 3 | 3 | 2 | 1 | 5 | 4 | 2 | 2 | 10 | 10 | 4 | 0 | 3 | 3 | 5 | 2 | 2 | 3 | 5 | 3
Cancer pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Catheter site related reaction (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Chills (General disorders) | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Facial pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Feeling cold (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
General physical health deterioration (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Irritability (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Localised Oedema (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oedema (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 1 | 0 | 0 | 2 | 0 | 0 | 1 | 1 | 0 | 1 | 2 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Pain (General disorders) | 1 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 1 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Puncture site haemorrhage (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Puncture site pain (General disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Puncture site reaction (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0 | 0 | 0 | 3 | 0 | 2 | 1 | 1 | 4 | 2 | 0 | 0 | 2 | 3 | 1 | 2 | 0 | 4 | 2
Sense of oppression (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Weight decreased (General disorders) | 1 | 0 | 2 | 0 | 1 | 2 | 4 | 4 | 3 | 5 | 2 | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 3 | 2
Weight increased (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Cholestasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cytolytic hepatitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Jaundice (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Anal abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aspergillosis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bacterial infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchopneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchopulmonary aspergillosis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Clostridial infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Device related infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Eye infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Folliculitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Fungal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gingival infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Herpes virus infection (Infections and infestations) | 0 | 0 | 1 | 2 | 1 | 0 | 1 | 2 | 2 | 3 | 2 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 1 | 1
Human herpesvirus 6 infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infection reactivation (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Localized infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lung infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Lyme disease (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lymphangitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oral candidiasis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oral fungal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Paronychia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Periodontal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Prostate infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Prostatitis escherichia coli (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory syncytial virus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rhinotracheitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tinea Cruris (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tonsillitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tooth abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Tooth infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tracheitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Viral skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vulvitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Excoriation (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eyelid injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Transfusion related complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aspergillus test positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bilirubin conjugated increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Blood magnesium decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
C-reactive protein increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Factor VII deficiency (Investigations) | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperbilirubinaemia (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
International normalised ratio (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
International normalised ratio decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
International normalised ratio increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0
Prothrombin time prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Prothrombin time shortened (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Transaminases increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 1 | 1 | 1 | 2 | 0 | 4 | 2 | 8 | 9 | 1 | 0 | 1 | 2 | 1 | 2 | 2 | 3 | 3 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Fluid overload (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fluid retention (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 0 | 3 | 4 | 3 | 0 | 3 | 5 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 3 | 0 | 3
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 0 | 1 | 2 | 1 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Obesity (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 2 | 0 | 0 | 1 | 0 | 2 | 1 | 0 | 2 | 0 | 0
Back disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 4 | 0 | 1 | 0 | 0 | 1 | 2 | 1 | 1 | 1 | 1
Bone disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle contracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 3 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 1 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Leukoerythroblastosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Anaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Balance disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Convulsion (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 2 | 4 | 0 | 1 | 0 | 0 | 2 | 1 | 3 | 0 | 4 | 1
Facial nerve disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 1 | 2 | 4 | 0 | 0 | 0 | 1 | 2 | 0 | 1 | 1 | 3 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Intracranial aneurysm (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Migraine (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Neuralgia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0
Peripheral motor neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Sinus headache (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Viith nerve paralysis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 0 | 2 | 1 | 0 | 1 | 1 | 3 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 5 | 1
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hallucination, visual (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Micturition urgency (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nocturia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Urinary hesitation (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract disorder (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract pain (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Breast pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nipple disorder (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Prostatitis (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chest pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 1 | 0 | 4 | 1 | 4 | 0 | 6 | 3 | 2 | 0 | 1 | 3 | 2 | 1 | 1 | 2 | 1 | 2
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 2 | 0 | 6 | 2 | 0 | 0 | 8 | 4 | 1 | 0 | 0 | 0 | 1 | 0 | 2 | 2 | 4 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 3 | 1 | 3 | 1 | 7 | 5 | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 1 | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Laryngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lung consolidation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis exfoliative (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1
Eccymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Erythrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 3 | 0
Intertrigo (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 4 | 2
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 1 | 0 | 2 | 0 | 1 | 1 | 1 | 0 | 2 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Purpura (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 5 | 2 | 1 | 0 | 1 | 0 | 2 | 1 | 0 | 1 | 2 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Scab (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Flushing (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 3 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hot flush (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 2 | 1
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Pallor (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Phlebitis (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thrombophlebitis superficial (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vasculitis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor has the opportunity to review all proposed publications regarding this trial 60 days prior to submission for publication. In addition, if requested, the investigator will withhold publication an additional 90 days to allow for filing a patent application or taking such other measures to establish and preserve its proprietary rights. Publication of the results of the study shall be made only as part of a publication of the results obtained by all sites performing the protocol.

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-03-10): https://cdn.clinicaltrials.gov/large-docs/82/NCT01713582/SAP_000.pdf
  • Study Protocol (2015-12-18): https://cdn.clinicaltrials.gov/large-docs/82/NCT01713582/Prot_001.pdf